CLINICAL TRIAL: NCT06996483
Title: Evaluation of the Effects of Oral Versus Intravenous 5-FU-Based Adjuvant Chemotherapy Regimens on Sleep Quality and Depression in Patients Diagnosed With Non-Metastatic Gastrointestinal System Cancer
Brief Title: Impact of Oral Versus Intravenous 5-FU-Based Adjuvant Regimens on Sleep Quality and Depression in Patients With Gastrointestinal Cancers
Acronym: FUSION
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncology, MD, Ankara Etlik City Hospital
Other Study IDs: AESH-EK1-2023-775
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Adjuvant Chemotherapy; 5-Fluorouracil; Sleep Quality; Depression; Gastrointestinal Cancer; Oral Chemotherapy; Intravenous Chemotherapy; Beck Depression Inventory; Pittsburgh Sleep Quality Index
MeSH Terms: conditions — Gastrointestinal Neoplasms; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral 5-FU Group: Patients receiving oral 5-FU-based adjuvant chemotherapy (e.g., capecitabine or CAPEOX) for non-metastatic gastrointestinal system cancers.
- Intravenous 5-FU Group: Patients receiving intravenous 5-FU-based adjuvant chemotherapy (e.g., FOLFOX) for non-metastatic gastrointestinal system cancers.

SUMMARY:
This prospective, non-randomized, single-center observational study is designed to investigate the effects of oral versus intravenous (IV) 5-fluorouracil (5-FU)-based adjuvant chemotherapy regimens on sleep quality and depression levels in patients with non-metastatic gastrointestinal system (GIS) cancers.

Eligible adult patients (aged 18 years or older) who are scheduled to receive adjuvant chemotherapy at the Ankara Etlik City Hospital Medical Oncology Department will be assessed using the Pittsburgh Sleep Quality Index (PSQI) and the Beck Depression Inventory (BDI). These evaluations will be conducted at baseline (prior to chemotherapy), on day forty-five, and on day ninety of treatment.

This study will not interfere with standard oncologic care. Instead, sleep disturbances and depressive symptoms will be monitored during routine clinical follow-up. Patients identified with significant psychological distress will be referred to psychiatry or sleep medicine departments for further evaluation.

The results of this study may provide insights into how different routes of 5-FU administration impact patients' mental health and quality of life, potentially informing future supportive care strategies during adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-center observational study designed to investigate the effects of oral versus intravenous (IV) 5-fluorouracil (5-FU)-based adjuvant chemotherapy regimens on sleep quality and depression levels in patients with non-metastatic gastrointestinal system (GIS) cancers.

The study will be conducted at the Ankara Etlik City Hospital, Medical Oncology Department. A total of 100 adult patients (≥18 years) who are initiating adjuvant chemotherapy including 5-FU (either oral or IV formulation) for histopathologically confirmed non-metastatic GIS cancers will be included.

Eligible patients will be enrolled after providing informed consent. The Pittsburgh Sleep Quality Index (PSQI) and Beck Depression Inventory (BDI), both of which have been validated in Turkish, will be used to assess sleep quality and depression severity. These measurements will be obtained at three time points: (1) baseline (prior to chemotherapy initiation), (2) day 45, and (3) day 90 of treatment.

The study aims to detect early psychosocial changes that may occur during chemotherapy, particularly those related to sleep and mood. No changes or interventions will be made to the patients' standard oncological treatment. Patients showing severe sleep disturbances or depressive symptoms during follow-up will be referred to the relevant departments (psychiatry or sleep medicine) for further evaluation and care.

The goal of the study is to better understand how the route of 5-FU administration (oral vs. IV) influences sleep patterns and emotional well-being during adjuvant chemotherapy. This could help optimize supportive care strategies and improve the quality of life of patients undergoing treatment for GIS cancers.

Data will be analyzed using appropriate statistical tests. Categorical variables will be compared using Chi-square or Fisher's exact test; continuous variables will be compared using Student's t-test or Mann-Whitney U test, depending on distribution. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed non-metastatic gastrointestinal system cancer (e.g., colorectal, gastric)
* Age ≥18 years
* Planned to receive adjuvant chemotherapy containing 5-FU (either oral or IV)
* ECOG performance status 0-2
* Provided informed consent

Exclusion Criteria:

* Patients with psychiatric disorders affecting sleep or mood
* Receiving treatment for primary sleep disorders or depression
* Prior chemotherapy or radiotherapy for the current diagnosis
* Inability to complete the questionnaires due to cognitive or language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-metastatic gastrointestinal cancers who are receiving adjuvant chemotherapy with oral or intravenous 5-fluorouracil-based regimens at a tertiary cancer center.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality Score (Pittsburgh Sleep Quality Index - PSQI) | Baseline, Day 45, Day 90
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) at Sleep quality will be assessed using the full version of the Pittsburgh Sleep Quality Index (PSQI) at three time points: prior to chemotherapy initiation (baseline), at day forty-five, and at day ninety.
  The PSQI total score ranges from 0 to 21, with higher scores indicating worse sleep quality. A score >5 is commonly used to define poor sleep quality.
  Changes over time within groups and differences between the oral 5-FU and intravenous 5-FU treatment groups will be analyzed.

SECONDARY OUTCOMES:
Change in Depression Score (Beck Depression Inventory - BDI) | Baseline, Day 45, Day 90
  Depression severity will be measured using the Beck Depression Inventory (BDI-I) at baseline, day forty-five, and day ninety.
  The BDI total score ranges from 0 to 63, with higher scores indicating more severe depressive symptoms.
  Standard interpretation categories are:
  0-13: minimal depression
  14-19: mild
  20-28: moderate
  29-63: severe
  Changes over time and comparisons between the oral and intravenous 5-FU groups will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Osman Sütcüoğlu, MD, Study Director — Etlik City Hospital, Medical Oncology Department
Locations (3):
- Turkey (Türkiye) (3):
  - Ankara Etlik City Hospital, Ankara, Yenimahalle
  - Etlik City Hospital, Medical Oncology Department, Ankara, Yenimahalle
  - Etlik City Hospital, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to local data protection regulations, ethical restrictions, and the absence of prior consent for data sharing.